CLINICAL TRIAL: NCT03814317
Title: An Open-Label Study of Inhaled Treprostinil in Sarcoidosis Patients With Pulmonary Hypertension and Interstitial Lung Disease (SAPPHIRE)
Brief Title: Inhaled Treprostinil in Sarcoidosis Patients With Pulmonary Hypertension
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCR19684; 20192572 (Other: WIRB)
Record Dates: First submitted 2019-01-04; First posted 2019-01-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Sarcoidosis; Precapillary Pulmonary Hypertension; Interstitial Lung Disease
Keywords: right heart catheterization (RHC); pulmonary vascular resistance (PVR); mean pulmonary arterial pressure (mPAP); pulmonary hypertension (PH); Inhaled treprostinil; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis; Lung Diseases, Interstitial; Hypertension, Pulmonary | interventions — treprostinil; hydralazine 4-anisaldehyde hydrazone; Therapeutics

STUDY DESIGN:
Intervention Model Description: All subjects will initiate inhaled treprostinil at a dose of 3 breaths (18 mcg) four times daily. Study drug doses escalations (additional one breath four times daily) can occur every three days with a maximum dosing regimen of up to 12 breaths (72 mcg) four times daily, as clinically tolerated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Sarcoidosis patients with interstitial lung disease and precapillary pulmonary hypertension based on right heart catheterization (RHC).
  All subjects will initiate inhaled treprostinil at a dose of 3 breaths (18 mcg) four times daily. Study drug doses escalations (additional one breath four times daily) can occur every three days with a maximum dosing regimen of up to 12 breaths (72 mcg) four times daily, as clinically tolerated.
  Interventions: Drug: Inhaled Treprostinil

INTERVENTIONS:
Drug: Inhaled Treprostinil — Inhaled treprostinil causes dilatation of the pulmonary arteries and may help reduce the pulmonary pressures in this studied population.
  All subjects will initiate inhaled treprostinil at a dose of 3 breaths (18 mcg) four times daily. Study drug doses escalations (additional one breath four times daily) can occur every three days with a maximum dosing regimen of up to 12 breaths (72 mcg) four times daily, as clinically tolerated.
  Other Names: Tyvaso®; pulmonary arterial hypertension (PAH) therapy

SUMMARY:
This study aims to evaluate the efficacy and safety of inhaled treprostinil in subjects with sarcoidosis-associated interstitial lung disease and pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary sarcoidosis-associated pulmonary hypertension is classified as WHO Group 5 pulmonary hypertension and may occur in anywhere from 5-20% of sarcoidosis patients. Inhaled treprostinil has shown clinical improvements in exercise capacity after 12 weeks of therapy in patients with WHO Group 1 pulmonary hypertension. More recently, there has been interest in using inhaled PAH-specific therapies for the treatment of pulmonary hypertension associated with interstitial lung disease.

The investigators believe that those patients with pulmonary hypertension in the setting of sarcoidosis-associated interstitial lung disease are a unique population which may potentially benefit from inhaled, targeted pulmonary arterial hypertension therapy (inhaled treprostinil) while minimizing the adverse effects associated with systemic pulmonary vasodilators. This study aims to evaluate the efficacy and safety of inhaled treprostinil in subjects with sarcoidosis-associated interstitial lung disease and pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Study participant willing and able to provide informed consent
* Negative urine pregnancy test at baseline for females of childbearing potential
* Established diagnosis of sarcoidosis by ATS/ERS/WASOG 1999 Statement on of Sarcoidosis
* Presence of interstitial lung disease by Scadding Stage IV chest radiograph or extensive fibrosis on chest computed tomography
* Right heart catheterization within six months of baseline visit showing precapillary pulmonary hypertension (mPAP ≥ 25 mmHg, PCWP ≤ 15 mmHg, and PVR > 3 WU)
* Patient on stable sarcoidosis therapy for at least three months prior to screening
* If patients are on oral PAH therapy (PDE5i/SCGS and/or ERA) then dose should be stable for at least three months prior to screening
* A 6MWT within three months of screening visit of > 100 meters

Exclusion Criteria:

* Pregnant patients or those who are actively lactating
* Patient not willing to use form of birth control (if applicable) during the study
* Inability to undergo 6MWT, RHC, PFTs or CMRI
* Predicted survival < 6 months
* Patient on any prostanoid or prostanoid analog therapy
* Patients with left sided heart disease as defined by either a PCWP > 15 mmHg and/or left ventricular ejection fraction < 40%
* Use of any investigational drug/device, or participation in any investigational study with therapeutic intent within 30 days prior to randomization.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
PVR by Right heart catheterization (RHC) | Baseline, Week 16
  Change in RHC parameter PVR (pulmonary vascular resistance )
mPAP by Right heart catheterization (RHC) | Baseline, Week 16
  Change in RHC parameter mPAP (mean pulmonary arterial pressure)

SECONDARY OUTCOMES:
Change in 6-Minute Walk Test (6MWT) | Baseline, Week 8, Week 16
  change in walk test distance during the study
Change in Cardiac MRI parameters | Baseline, Week 16
  Change in Right ventricle ejection fraction, Right ventricular end diastolic ventricle index, right ventricular systolic index
Change in Pulmonary Function Testing | Baseline, Week 16
  Change in FEV1 abd FVC
Change in Brain Natriuretic Peptide (BNP) | Baseline, Week 16
  change in BNP level during the study
Change in WHO Functional Class (WHO FC) | Baseline, Week 8, Week 16
  change in WHO FC status during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ataya, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Division of Pulmonary and Critical Care Medicine, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No